CLINICAL TRIAL: NCT07284173
Title: A Phase 1, Open Label, Fixed Sequence Study to Investigate the Effect of Rabeprazole on the Pharmacokinetics of PF-08049820 in Healthy Chinese Adult Participants.
Brief Title: A Study to Learn if a Medicine That Reduces Stomach Acid Affects the Blood Level of Study Medicine PF-08049820 in Healthy Chinese Adults.
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Basic Science
Other Study IDs: C6231005
Record Dates: First submitted 2025-11-13; First posted 2025-12-16 (Actual); Last update posted 2025-12-16 (Actual); Status verified 2025-12

CONDITIONS: Healthy Adults
Keywords: Healthy; Atopic Dermatitis
MeSH Terms: conditions — Dermatitis, Atopic | interventions — Rabeprazole

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Treatment A (Experimental): Participants will receive single oral dose of PF-08049820.
  Interventions: Drug: PF-08049820
- Treatment B (Experimental): Participants will receive rabeprazole for 5 days followed by a single oral dose of PF-08049820 and rabeprazole.
  Interventions: Drug: PF-08049820; Drug: Rabeprazole

INTERVENTIONS:
Drug: PF-08049820 — Oral tablets
Drug: Rabeprazole — Oral tablets
  Other Names: Pariet
  Arms: Treatment B

SUMMARY:
This clinical study is designed to evaluate a study medicine called PF-08049820. The main aim is to understand how the body processes this medicine and whether giving it with another medicine, rabeprazole, affects how it behaves.

The study will take in healthy adult participants aged 18 to 65 years who are not able to have children. Eligible participants must weigh more than 50 kilograms (110 pounds) and have a Body Mass Index (BMI) between 18.5 and 27.9.

Each participant will receive two treatments:

* One treatment with PF-08049820 alone
* One treatment with PF-08049820 taken together with rabeprazole

Both medicines will be taken by mouth. Participants will stay at the study clinic for a few days during each treatment period. During these stays, the study team will collect blood samples to see how the body absorbs and processes the medicine.

ELIGIBILITY:
Inclusion Criteria:

* Male and female participants of non-childbearing potential aged 18 to 65 years, inclusive, at screening who are overtly healthy as determined by medical evaluation including medical history, physical examination, laboratory tests, and 12-lead electrocardiogram.
* BMI of 18.5-27.9 kg/m2; and a total body weight >50 kg (110 lb).
* Participants who are willing and able to comply with all scheduled visits, treatment plans, laboratory tests, and other study procedures.

Exclusion Criteria:

* History or evidence of significant hematological, renal, endocrine, pulmonary, gastrointestinal, cardiovascular, hepatic, psychiatric, neurological, or allergic diseases.
* Positive test for HIV, hepatitis B (HBsAg), or hepatitis C (HCVAb).
* Active or latent tuberculosis (TB) infection or inadequate treatment history for TB.
* Any medical or psychiatric condition, including active suicidal ideation in the past year or suicidal behavior in the past 5 years, that may increase risk or interfere with study participation.
* Current use of prohibited medications or inability/unwillingness to use required medications.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2025-11-03 (Actual); Primary Completion 2025-12-15 (Estimated); Study Completion 2025-12-15 (Estimated)

PRIMARY OUTCOMES:
Pharmacokinetics (PK): Maximum Observed Plasma Concentration (Cmax) of PF-08049820. | Day 1 through Day 38-45
PK: Area under the plasma concentration (AUC) of PF-08049820 | Day 1 through Day 38-45

SECONDARY OUTCOMES:
Number of participants with treatment emergent adverse events | First dose through Day 38-45

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Beijing Friendship Hospital Affiliate of Capital University, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=C6231005